CLINICAL TRIAL: NCT05958472
Title: Study on Glioma Patients: Understanding Their Glioma Clinical Trial Experiences
Brief Title: Navigating the Clinical Research Process for Glioma
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81932689
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Glioma
Keywords: glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in medical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This trial will admit a wide range of data on the clinical trial experience of glioma patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future glioma patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of glioma
* Participant must be 18 years of age or older
* Participant must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study.

Exclusion Criteria:

* Pregnant or lactating woman
* Participant is actively receiving study therapy in another
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioma patients who are actively considering participating in a clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a glioma clinical research. | 3 months
Number of glioma study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Meer PB, Dirven L, Fiocco M, Vos MJ, Kouwenhoven MCM, van den Bent MJ, Taphoorn MJB, Koekkoek JAF. Effectiveness of Antiseizure Medication Duotherapies in Patients With Glioma: A Multicenter Observational Cohort Study. Neurology. 2022 Sep 6;99(10):e999-e1008. doi: 10.1212/WNL.0000000000200807. Epub 2022 Jun 8. PMID 36219797
- [Background] Epstein RH, Dexter F, Cajigas I, Mahavadi AK, Shah AH, Abitbol N, Komotar RJ. Prolonged tracheal extubation time after glioma surgery was associated with lack of familiarity between the anesthesia provider and the operating neurosurgeon. A retrospective, observational study. J Clin Anesth. 2020 Mar;60:118-124. doi: 10.1016/j.jclinane.2019.09.003. Epub 2019 Oct 24. PMID 31669746
- [Background] Berntsson SG, Merrell RT, Amirian ES, Armstrong GN, Lachance D, Smits A, Zhou R, Jacobs DI, Wrensch MR, Olson SH, Il'yasova D, Claus EB, Barnholtz-Sloan JS, Schildkraut J, Sadetzki S, Johansen C, Houlston RS, Jenkins RB, Bernstein JL, Lai R, Shete S, Amos CI, Bondy ML, Melin BS. Glioma-related seizures in relation to histopathological subtypes: a report from the glioma international case-control study. J Neurol. 2018 Jun;265(6):1432-1442. doi: 10.1007/s00415-018-8857-0. Epub 2018 Apr 23. PMID 29687214

DOCUMENTS (1):
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT05958472/ICF_000.pdf